CLINICAL TRIAL: NCT03527862
Title: The Effect of Perioperative Lung Ultrasonography on Postoperative Outcomes in Children Undergoing Fast-track Cardiac Surgery
Brief Title: Perioperative Lung Ultrasonography for Fast-track Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H1803-123-932
Record Dates: First submitted 2018-04-24; First posted 2018-05-17 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No intervention is performed. Lung ultrasonography is performed within 4 hours after surgery for diagnostic purpose.
- lung ultrasonography group (Experimental): Lung ultrasonography is performed three times; after tracheal intubation, before surgery end, and within 4 hours after surgery. In this group, respiratory management is performed according to diagnosis.
  Interventions: Other: Treatment according to lung ultrasonography

INTERVENTIONS:
Other: Treatment according to lung ultrasonography — Appropriate treatment for atelectasis, pleural effusion, pulmonary edema, pneumothorax or pneumonia which are confirmed by lung ultrasonography
  Arms: lung ultrasonography group

SUMMARY:
The investigators evaluate the usefulness of lung ultrasonography in the perioperative period for postoperative outcomes in children undergoing fast track cardiac surgery.

DETAILED DESCRIPTION:
Some appropriate intervention such as recruitment maneuver, chest tube insertion, or diuretics will be applied depending on lung ultrasound findings.

ELIGIBILITY:
Inclusion Criteria:

* Children receiving fast track cardiac surgery protocol
* = or < 5 years old
* Children with acyanotic heart disease

Exclusion Criteria:

* Previous history of lung resection surgery
* Preoperative chest x-ray abnormalities
* Postoperative cyanosis

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2018-05-08 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | Up to postoperative day 5
  Pleural effusion, atelectasis, diaphragmatic dysfunction, pulmonary infection, embolism, respiratory failure, aspiration, pneumothorax, chylothorax, bronchospasm

SECONDARY OUTCOMES:
Duration of the use of inotropes | Up to postoperative day 5
  Duration of the use of inotropes
Length of intensive care unit stay | up to postoperative day 5
  Length of intensive care unit stay
Lung ultrasonography findings | until 4 hours after surgery
  Diagnostic lung ultrasonography
ABGA result | within 4 hours after extubation
  arterial blood gas analysis results
Duration of oxygen therapy | Up to postoperative day 5

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea